CLINICAL TRIAL: NCT01888432
Title: A 24 Month, Randomized, Controlled, Study to Evaluate the Efficacy and Safety of Concentration-controlled Everolimus Plus Reduced Tacrolimus Compared to Standard Tacrolimus in Recipients of Living Donor Liver Transplants and Long Term Extension to Evaluate the Efficacy and Safety of Concentration-controlled Everolimus Plus Reduced Tacrolimus Compared to Standard Tacrolimus in Recipients of Living Donor Liver Transplants in Japan
Brief Title: Efficacy and Safety of Everolimus in Liver Transplant Recipients of Living Donor Liver Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRAD001H2307; 2010-024527-25 (EudraCT Number)
Record Dates: First submitted 2013-06-15; First posted 2013-06-27 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-02

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; everolimus; tacrolimus; reduced calcineuron inhibitor; renal function; living donor; RAD001H2307; RAD001H
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Intervention Model Description: This was a 24-month, multicenter, open-label, randomized, controlled study. It included the extension to the 24-month, randomized, controlled, open-label CRAD001H2307 study in recipients of living donor liver transplants in Japan.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Everolimus + reduced tacrolimus (Experimental): Everolimus + reduced tacrolimus ± corticosteroids
  Interventions: Drug: Everolimus + reduced tacrolimus
- Standard tacrolimus (Active Comparator): Standard tacrolimus ± corticosteroids
  Interventions: Drug: Standard tacrolimus

INTERVENTIONS:
Drug: Everolimus + reduced tacrolimus — Everolimus was initiated at Week 4 post transplantation. The dose was adjusted to maintain the everolimus trough blood levels between 3-8 ng/mL for the duration of the study. Tacrolimus was reduced to 3-5 ng/mL.
  Arms: Everolimus + reduced tacrolimus
Drug: Standard tacrolimus — Tacrolimus was initiated as soon as possible after transplantation according to approved labeling recommendations. The trough level should've been 5-15 ng/mL until randomization, 8-12 ng/mL from randomization until month 4 and after month 4 until end of study reduced to 6 -10 ng/mL.
  Arms: Standard tacrolimus

SUMMARY:
The purpose of this trial was to demonstrate the efficacy and safety of everolimus in combination with reduced tacrolimus, compared to tacrolimus control, in living donor liver transplant recipients.

DETAILED DESCRIPTION:
This study was 24 month, multicenter study in 280 living donor liver transplant patients from Asia, Europe and Canada. The study has an long term extension in Japan and approximately 28 patients were to be included to evaluate the long-term efficacy and safety of concentration-controlled everolimus regimen plus reduced tacrolimus compared to standard tacrolimus in recipients of living donor liver transplants in Japan who participated in the CRAD001H2307 study.

Data reported here are the CRAD001H2307 core study results and its extension (CRAD001H2307E1).

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Subject aged ≥18 years of a primary, orthotopic liver allograft, from a living donor
* Subject negative for HIV

Incusion criteria at Randomization:

- Subject was initated on tacrolimus-based immunosuppressive regimen with steroids and other immunosuppression

Exclusion criteria:

* Subjects transplanted for acute liver failure
* HCV negativesubjects receiving a transplant from HCV positive donor
* Subjects receiving multiple solid organ (including multiple liver lobes/segments) or islet cell tissue transplants, or have previously received an organ or tissue transplant.
* Subjects receiving an ABO incompatible allograft.
* MELD-score > 35 within 1 month prior to transplantation.
* Use of immunosuppressive or antibody induction agents not specified in the protocol.
* History of malignancy of any organ system (except hepatocellular carcinoma or localized basal cell carcinoma of the skin)
* Hepatocellular carcinoma with extrahepatic spread or macrovascular invasion
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 2 weeks after the last dose of study medication
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical class, or to any of the excipients

Exclusion criteria at Randomization:

* Any post-transplant history of thrombosis, occlusion or stent placement in any major hepatic arteries, hepatic veins, portal vein or inferior vena cava at any time during the run-in period prior to randomization.
* Subjects with a confirmed spot urine protein/creatinine ratio that indicates ≥ 1.0 g/24 hrs of proteinuria
* Subjects who have severe hypercholesterolemia (>350 mg/dL; >9.1 mmol/L) or hypertriglyceridemia (>500 mg/dL; >5.6 mmol/L) at randomization.
* Subjects with platelet count < 30,000/mm3.
* Subjects with an absolute neutrophil count of < 1,000/mm³ or white blood cell count of < 2,000/mm³.
* Subjects with systemic infection requiring active use of IV antibiotics.
* Subjects requiring life support measures such as ventilation, dialysis, vasopressor agents.
* Subjects who require renal replacement therapy within 7 days prior to randomization.
* Subjects with detectable HBV DNA at time of randomization
* Subjects meeting the following criteria for acute rejection during the run in period:

  * Any acute rejection in the week prior to randomization.
  * 2 treated acute rejections.
  * Any rejection requiring antibody treatment.
  * Any severe cellular (and/or any humoral) rejection.

Long term extension for patients in Japan:

Inclusion criteria

* Written informed consent must be obtained before any extension specific assessment is performed.
* Ability and willingness to adhere to study regimen.
* Completed Month 24 visit of core study and continuously being treated with assigned regimen.

Exclusion criteria:

* Use of medication that is prohibited by the study protocol at Month 24.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical class, or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2018-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- United States (9):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlottesville, Virginia
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Cairo, Egypt
- Germany (4):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
- India (3):
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Chennai, Tamil Nadu
- Novartis Investigative Site, Milan, MI, Italy
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sakyo Ku, Kyoto
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Seoul, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Malatya
  - Novartis Investigative Site, Mecidiyekoy/Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Jeng LB, Lee SG, Soin AS, Lee WC, Suh KS, Joo DJ, Uemoto S, Joh J, Yoshizumi T, Yang HR, Song GW, Lopez P, Kochuparampil J, Sips C, Kaneko S, Levy G. Efficacy and safety of everolimus with reduced tacrolimus in living-donor liver transplant recipients: 12-month results of a randomized multicenter study. Am J Transplant. 2018 Jun;18(6):1435-1446. doi: 10.1111/ajt.14623. Epub 2018 Jan 25. PMID 29237235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In all, 284 patients were randomized after transplantation to EVR+Reduced TAC group and TAC Control group. Two patients were not eligible and randomized in IRT by mistake and to whom no study medication was given, and so did not have their data included.
Pre-assignment Details: A total of 494 patients were screened. Of these, 448 patients received a liver transplant and entered the run-in period.
Groups:
- EVR+Reduced TAC: Everolimus + reduced tacrolimus ± corticosteroids
- TAC Control: Standard tacrolimus ± corticosteroids
Period: 12-month Analysis (FAS)
Arm/Group | EVR+Reduced TAC | TAC Control
Started | 142 | 142
Completed | 131 | 133
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Death | 4 | 3
Period: 24-month Analysis (FAS)
Arm/Group | EVR+Reduced TAC | TAC Control
Started | 142 | 142
Completed | 125 | 125
Not Completed | 17 | 17
Not completed — Graft loss | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 2 | 4
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Death | 8 | 4
Period: 36-month Analysis (Extension)
Arm/Group | EVR+Reduced TAC | TAC Control
Started | 13 | 5
Completed | 12 | 5
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): patients were analyzed according to treatment assigned at randomization. Any subject without written informed consent signed did not have their data included. Mis-randomized patients, who were not eligible but randomized in IRT by mistake and to whom no study medication was given, did not have their data included.
Groups:
- Total: Total of all reporting groups
Arm/Group | EVR+Reduced TAC | TAC Control | Total
Number analyzed (Participants) | 142 | 142 | 284
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (8.95) | 52.7 (10.41) | 53.5 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 43 | 81
  Male | 104 | 99 | 203
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 30 | 30 | 60
  Asian | 111 | 112 | 223
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Efficacy Failure of Treated Biopsy Proven Acute Rejection, Graft Loss or Death in Everolimus With Reduced Tacrolimus Group Compared to Standard Tacrolimus
Description: Rate of composite efficacy failure of treated biopsy proven acute rejection (tBPAR ≥ RAI score 3), graft loss (GL) or death (D) in everolimus with reduced tacrolimus group compared to standard tacrolimus at 12 months
Time Frame: 12 months post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants | 7 | 8
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; non-inferior efficacy failure of the reduced tacrolimus regimen to control by rejecting the null hypothesis; Test type: Non-Inferiority — HO: πT - πC ≥ 0.12 vs. HA: πT - πC < 0.12, where πT and πC are the true proportions of composite efficacy failure of tBPAR, GL, or D, (tBPAR/GL/D) at 12 months post-transplant for the respective treatment groups. The proportion of 0.12, or 12%, was pre-determined as the non-inferiority (NI) margin for composite efficacy failure; p < 0.001, Z-test — Z-test p-value for non-inferiority test (non-inferiority margin = 12%) is for one-sided test and should be compared to 0.05 significance level; Kaplan-Meier = -0.7, 90% CI 2-sided [-5.2 to 3.7]

2. Secondary Outcome: Renal Function by Estimated Glomerular Filtration Rate (eGFR) From Randomization
Description: Renal function (change in estimated glomerular filtration rate (eGFR)) from randomization to Month 12 post transplantation with everolimus (EVR) in combination with reduced tacrolimus (rTAC) compared to standard exposure tacrolimus (TAC) in living donor liver transplant recipients.
Time Frame: From randomization to month 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
mL/min/1.73 m^2 | -7.94 (1.839) | -12.09 (1.824)
Statistical Analysis 1: Comparison: EVR+Reduced TAC; Test type: Non-Inferiority — the null hypothesis below was tested at the one-sided α = 0.05 level: H0: μT - μC ≤ -6 mL/min/1.73 m2 vs. HA: μT - μC > -6 mL/min/1.73 m^2, where μT and μC are the true means of change in eGFR (MDRD-4) from randomization to Month 12 post-transplant for the reduced tacrolimus group and control group, respectively; p < 0.001, ANCOVA; Mean Difference (Net) = 4.15, 90% CI 2-sided [-0.09 to 8.40], Standard Error of Mean 2.574

3. Secondary Outcome: Compare Renal Function Over Time Assessed by the Change by eGFR, Post-randomization
Description: Change in renal function from randomization to month 24 assessed by the change in estimated GFR (MDRD-4). Rate of change of renal function.
Time Frame: From randomziation to month 24
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m2
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
mL/min/1.73 m2 | -11.01 (1.928) | -14.26 (1.914)
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.25, 90% CI 2-sided [-1.21 to 7.70], Standard Error of Mean 2.699

4. Secondary Outcome: Number of Participants With Composite of tBPAR, Graft Loss, and Death
Description: Compare between the treatment group EVR with rTAC vs standard TAC: incidence of a composite of tBPAR, graft loss, death
Time Frame: Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  tBPAR/graft loss/death | 12 | 11
  On-treatment tBPAR/graft loss/death | 7 | 9

5. Secondary Outcome: Compare Incidence of tBPAR
Description: Compare between the treatment group EVR with rTAC vs standard TAC: Incidence of tBPAR
Time Frame: Month 12 and Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  tBPAR - month 12 | 3 | 5
  tBPAR - month 24 | 4 | 6
  On-treatment tBPAR - month 24 | 3 | 6
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 12; Kaplan-Meier = -1.4, 90% CI 2-sided [-4.7 to 2.0] — KM rate and 90% CI are obtained using KM probability estimates of composite efficacy failure rates and standard error derived based on Greenwood's formula
Statistical Analysis 2: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — tBPAR - month 24; Kaplan-Meier = -1.2, 90% CI 2-sided [-5.1 to 2.6] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — On-treatment tBPAR - month 24; Kaplan-Meier = -2.1, 90% CI 2-sided [-5.7 to 1.4] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Compare Incidence of BPAR
Description: Compare between the treatment group EVR with rTAC vs standard TAC: incidence of a composite of biopsy proven acute rejection (BPAR)
Time Frame: Month 12 and Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  Month 12 | 7 | 6
  Month 24 | 8 | 7
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 12; Kaplan-Meier = 0.9, 90% CI 2-sided [-3.4 to 5.1] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 24; Kaplan-Meier = 1.0, 90% CI 2-sided [-3.6 to 5.6] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Compare Incidence of Graft Loss
Description: Compare between the treatment group EVR with rTAC vs standard TAC: incidence of graft loss
Time Frame: Month 12 and Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  Month 12 | 0 | 0
  month 24 | 0 | 1
  month 24 (on-treatment graft loss) | 0 | 0
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — graft loss at month 24; Kaplan-Meier = -0.8, 90% CI 2-sided [-2.1 to 0.5] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Compare Incidence of a Composite of Death or Graft Loss
Description: Compare between the treatment group EVR with rTAC vs standard TAC: Incidence of a composite of death or graft loss
Time Frame: Month 12 and Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  Month 12 | 4 | 3
  Month 24 | 8 | 5
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 12; Kaplan-Meier = 0.7, 90% CI 2-sided [-2.5 to 3.8] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 24; Kaplan-Meier = 2.3, 90% CI 2-sided [-2.1 to 6.6] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Compare Incidence of Death
Description: Compare between the treatment group EVR with rTAC vs standard TAC: incidence of death
Time Frame: Month 12 and Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  Month 12 | 4 | 3
  Month 24 | 8 | 4
  Month 24 (on-treatment death) | 4 | 3
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 12; Kaplan-Meier = 0.7, 90% CI 2-sided [-2.5 to 3.8] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 24; Kaplan-Meier = 3.0, 90% CI 2-sided [-1.1 to 7.2] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other — Month 24 (On-treatment death); Kaplan-Meier = 0.7, 90% CI 2-sided [-2.5 to 3.9] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Compare Incidence of AR
Description: Compare between the treatment group EVR with rTAC vs standard TAC: incidence of acute rejection (AR)
Time Frame: Month 12 and Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  Month 12 | 9 | 8
  Month 24 | 12 | 9
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Risk Difference (RD) = 0.7, 90% CI 2-sided [-3.9 to 5.3] — Month 12
Statistical Analysis 2: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Risk Difference (RD) = 2.1, 90% CI 2-sided [-3.0 to 7.2] — Month 24

11. Secondary Outcome: Compare Incidence of tAR
Description: Compare between the treatment group EVR with rTAC vs standard TAC: incidence of treated acute rejection (tAR).
Time Frame: Month 12 and Month 24 post transplantation
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 142
Participants
  Month 12 | 5 | 6
  Month 24 | 7 | 7
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Risk Ratio (RR) = -0.7, 90% CI 2-sided [-4.5 to 3.1] — Month 12
Statistical Analysis 2: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Risk Ratio (RR) = 0.0, 90% CI 2-sided [-4.2 to 4.2] — Month 24

12. Secondary Outcome: Number of Participants With Time to Recurrence of HCC in Subjects With a Diagnosis of HCC at the Time of Liver Transplantation
Description: Patients transplanted for HCC or with HCC diagnosed at time of transplantation were monitored for HCC recurrence according to local practice. For example routine laboratory monitoring/tests, tumor markers, hepatic ultrasound, computed tomography scans (CAT, CT) or MRI (especially Fe-MRI) on a regular basis per local practice.
Time Frame: Month 12 and Month 24
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 141
Participants
  HCC recurrence (n/M) - month 12: number analyzed (Participants) | 56 | 62
  HCC recurrence (n/M) - month 12 | 0 | 5
  HCC recurrence (n/M) - month 24: number analyzed (Participants) | 56 | 61
  HCC recurrence (n/M) - month 24 | 1 | 6

13. Secondary Outcome: Number of Subjects Experiencing Adverse Events/Infections by SOC
Time Frame: Month 24
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 141
Participants
  Any AE/infection | 140 | 136
  Blood and lymphatic system disorders | 44 | 32
  Cardiac disorders | 15 | 12
  Congenital, familial and genetic disorders | 1 | 2
  Ear and labyrinth disorders | 2 | 5
  Endocrine disorders | 1 | 2
  Eye disorders | 17 | 15
  Gastrointestinal disorders | 98 | 74
  General disorders&admin site conditions | 48 | 42
  Hepatobiliary disorders | 44 | 40
  Immune system disorders | 8 | 11
  Infections and infestations | 84 | 70
  Injury, poisoning&proced. complications | 36 | 28
  Investigations | 61 | 68
  Metabolism and nutrition disorders | 87 | 60
  Musculoskeletal and connective tissue disorders | 30 | 43
  Neoplasms benign, malig&unspecified (cysts&polyps) | 10 | 17
  Nervous system disorders | 38 | 44
  Product issues# | 1 | 1
  Psychiatric disorders | 33 | 26
  Renal and urinary disorders | 46 | 36
  Reproductive system&breast dis. | 9 | 12
  Respiratory, thoracic&mediastinal dis. | 34 | 39
  Skin&subcutaneous tissue disorders | 39 | 44
  Vascular disorders | 38 | 30

14. Secondary Outcome: Compare Incidence of Notable Safety Events (SAEs, Infections and Serious Infections Leading to Premature Discontinuation)
Description: Notable events include death, Serious AE/infection,, and AE/infection leading to discontinuation of study medication.
Time Frame: Month 24
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 142 | 141
Participants
  Any notable events | 86 | 82
  Death | 8 | 4
  Serious AE/Infection | 83 | 78
  AE/Infection lead. to premature disc of study med | 21 | 18

15. Secondary Outcome: Composite Efficacy Failure of Treated Biopsy in Everolimus With Reduced Tacrolimus Group Compared to Standard Tacrolimus in Patients From Japan Only
Description: Rate of composite efficacy failure of treated biopsy in everolimus with reduced tacrolimus group compared to standard tacrolimus from randomization in core study up to 36 months in the extension study.
  Composite endpoint = treated BPAR, graft loss or death. AR = Acute rejection; tAR = treated AR; BPR = biopsy proven rejection; BPAR = biopsy proven acute rejection; tBPAR = treated BPAR
Time Frame: randomization, 36 months post transplantion
Population: All extension patients consisted of all patients enrolled into this extension study.
Measure: Number; unit: Participants
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 16 | 12
Participants
  Composite endpoint | 2 | 1
  On-treatment composite endpoint | 1 | 0
  Graft loss/death | 1 | 1
  tBPAR | 2 | 0
  Graft loss | 0 | 1
  Death | 1 | 0
  AR | 3 | 2
  tAR | 2 | 0
  BPR | 6 | 3
  BPAR | 3 | 2
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 5.4, 95% CI 2-sided [-19.9 to 30.6] — Composite endpoint
Statistical Analysis 2: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 6.7, 95% CI 2-sided [-6.0 to 19.3] — On-treatment composite endpoint
Statistical Analysis 3: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 2.0, 95% CI 2-sided [-24.6 to 28.7] — Graft loss/death
Statistical Analysis 4: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 14.4, 95% CI 2-sided [-4.2 to 33.1] — tBPAR
Statistical Analysis 5: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 11.1, 95% CI 2-sided [-9.4 to 31.6] — Death
Statistical Analysis 6: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 3.2, 95% CI 2-sided [-28.9 to 35.2] — AR
Statistical Analysis 7: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 14.4, 95% CI 2-sided [-4.2 to 33.1] — tAR
Statistical Analysis 8: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 14.9, 95% CI 2-sided [-22.3 to 52.1] — BPR
Statistical Analysis 9: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Difference in Kaplan-Meier estimate = 3.2, 95% CI 2-sided [-28.9 to 35.2] — BPAR

16. Secondary Outcome: Renal Function by Estimated Glomerular Filtration Rate (All Extension Patients)
Description: Renal function (change in estimated glomerular filtration rate (eGFR)) from randomization to Month 36 post transplantation with everolimus (EVR) in combination with reduced tacrolimus (rTAC) compared to standard exposure tacrolimus (TAC) in living donor liver transplant recipients in Japan
Time Frame: randomization, at 36 months post transplantation
Population: All extension patients consisted of all patients enrolled into this extension study.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m2
Arm/Group | EVR+Reduced TAC | TAC Control
Number analyzed (Participants) | 13 | 5
mL/min/1.73m2 | -26.88 (10.114) | -16.87 (19.412)
Statistical Analysis 1: Comparison: EVR+Reduced TAC vs TAC Control; Test type: Other; Mean Difference (Final Values) = -10.01, 95% CI 2-sided [-59.91 to 39.89], Standard Error of Mean 22.059

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 4 years
Groups:
- AE From Day 1 to Month 24_EVR+Reduced TAC; AE From Month 24 to Month 36_EVR+Reduced TAC: Everolimus + reduced tacrolimus ± corticosteroids
- AE From Day 1 to Month 24_TAC Control; AE From Month 24 to Month 36_TAC Control: Standard tacrolimus ± corticosteroids
Arm/Group | AE From Day 1 to Month 24_EVR+Reduced TAC | AE From Day 1 to Month 24_TAC Control | AE From Month 24 to Month 36_EVR+Reduced TAC | AE From Month 24 to Month 36_TAC Control
All-Cause Mortality (participants affected / at risk) | 8/142 | 4/141 | 1/13 | 0/5
Serious Adverse Events (participants affected / at risk) | 83/142 | 78/141 | 5/13 | 0/5
Other Adverse Events (participants affected / at risk) | 127/142 | 122/141 | 13/13 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AE From Day 1 to Month 24_EVR+Reduced TAC (N=142) | AE From Day 1 to Month 24_TAC Control (N=141) | AE From Month 24 to Month 36_EVR+Reduced TAC (N=13) | AE From Month 24 to Month 36_TAC Control (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac discomfort (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0
Lens dislocation (Eye disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mesenteric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pouchitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestine ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Crepitations (General disorders) | 0 | 1 | 0 | 0
Hyperpyrexia (General disorders) | 1 | 0 | 0 | 0
Incarcerated hernia (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 11 | 8 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 10 | 6 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary fistula (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Biloma (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 8 | 9 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Portal vein stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Primary biliary cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver transplant rejection (Immune system disorders) | 3 | 3 | 0 | 0
Transplant rejection (Immune system disorders) | 2 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Arteriovenous graft site infection (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 2 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 0 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0
Fungal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 5 | 3 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 2 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 5 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Prostatic abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Graft loss (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 5 | 1 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 0
Hepatic enzyme increased (Investigations) | 4 | 2 | 0 | 0
Immunosuppressant drug level increased (Investigations) | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 1 | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bone giant cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 0
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Wernicke's encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Lymphangiopathy (Vascular disorders) | 0 | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Venous stenosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AE From Day 1 to Month 24_EVR+Reduced TAC (N=142) | AE From Day 1 to Month 24_TAC Control (N=141) | AE From Month 24 to Month 36_EVR+Reduced TAC (N=13) | AE From Month 24 to Month 36_TAC Control (N=5)
Anaemia (Blood and lymphatic system disorders) | 18 | 15 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 16 | 7 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 3 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 8 | 4 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 19 | 12 | 0 | 0
Anal erosion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 13 | 16 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 32 | 19 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 17 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 9 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 19 | 5 | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 10 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 16 | 8 | 1 | 0
Pyrexia (General disorders) | 18 | 20 | 3 | 1
Hepatic steatosis (Hepatobiliary disorders) | 10 | 7 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 6 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 2 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 1 | 0
Influenza (Infections and infestations) | 3 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 20 | 16 | 5 | 3
Pharyngitis (Infections and infestations) | 1 | 2 | 2 | 0
Pneumonia (Infections and infestations) | 4 | 2 | 2 | 0
Sepsis (Infections and infestations) | 4 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 18 | 11 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 8 | 2 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 2 | 6 | 0 | 1
Alanine aminotransferase increased (Investigations) | 5 | 8 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 6 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 1 | 0
Blood creatinine increased (Investigations) | 10 | 13 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 5 | 1 | 0
Hepatic enzyme abnormal (Investigations) | 8 | 19 | 0 | 0
Hepatic enzyme increased (Investigations) | 16 | 19 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 13 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 13 | 4 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 22 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 20 | 13 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 22 | 8 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 8 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 11 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 9 | 0 | 0
Headache (Nervous system disorders) | 19 | 14 | 1 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 4 | 11 | 0 | 0
Depression (Psychiatric disorders) | 2 | 8 | 0 | 0
Insomnia (Psychiatric disorders) | 26 | 13 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 4 | 6 | 1 | 0
Proteinuria (Renal and urinary disorders) | 6 | 2 | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 13 | 0 | 0
Renal impairment (Renal and urinary disorders) | 11 | 5 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 15 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 18 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 10 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Hypertension (Vascular disorders) | 29 | 23 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.